CLINICAL TRIAL: NCT03011008
Title: Effect of Liraglutide as Additional Treatment to Insulin in Patients With Autoimmune Diabetes Mellitus
Brief Title: Liraglutide as Additional Treatment to Insulin in Patients With Autoimmune Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Principal Investigator, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0002
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes Mellitus; Autoimmune Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide; Insulin

ARMS (2):
- Liraglutide + insulin (Experimental): Patients will be subjected to a dose escalation of liraglutide up to 1.2 mg, then continue to receive the reached liraglutide dose once daily for 6 months thereafter. Insulin will be continued as routine therapy.
  Interventions: Drug: Liraglutide; Drug: Insulin
- Insulin (Active Comparator): Patients will receive insulin injection as a routine therapy.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Liraglutide — Dose escalation of liraglutide starts from 0.6 mg up to 1.2 mg per day.
  Arms: Liraglutide + insulin
Drug: Insulin — Receive insulin following clinician's instruction.

SUMMARY:
The purpose of this study is to investigate the therapeutic effect of Liraglutide on autoimmune diabetes.

DETAILED DESCRIPTION:
Autoimmune Diabetes Mellitus (AIDM) is a subtype of diabetes mellitus caused by autoimmune destruction of beta cells in the islet, including Type 1 diabetes and Latent Autoimmune Diabetes in Adults (LADA). Insulin has been used as a routine therapy for AIDM to alleviate the hyperglycemic status, yet cannot effectively prevent the progressing destruction of beta cells or preserve its function. Glucagon-like peptide (GLP-1) analog Liraglutide has been tested in large-scale clinical trial to prove its various benefits for beta cells and glucolipid metabolism in Type 2 diabetes and obesity patients. However, its clinical application in AIDM is not well-defined so far. The aim of this study is to investigate the potential use of Liraglutide on glycemic control in AIDM.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes according to ADA criteria <3 years.
* Age≥ 18 years.
* Positive for at least one of the anti-islet autoantibodies: GADA, IA2A, ZnT8A
* Fasting or postprandial plasma C-peptide more than 100 pmol/L
* Written informed consent from the patient or family representative

Exclusion Criteria:

* History or family history of medullary thyroid carcinoma or MEN 2 syndrome;
* History of chronic or acute pancreatitis;
* Allergic to liraglutide or any components in Victoza®;
* Hepatic abnormalities (transaminase > 2 times normal);
* Renal impairments (serum creatinine >133 umol/L);
* Cardiovascular diseases (hypertension, coronary heart disease, etc.);
* Presence of acute metabolic disorders; In the case of acute ketone acidosis, with blood ketone over 0.3mmol/L and pH lower than 7.30;
* Any history of malignancy;
* Female patients who are pregnant or breastfeeding; any female who is unwilling to use a reliable and effective form of contraception for 2 years after recruitment;
* Presence of any infectious diseases, including active skin infections, flu, fever, upper or lower respiratory tract infections; those who wish to participate in the study should keep the infection under control for at least 1 week before receiving Treg product infusion;
* Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Mean amplitude of glycemic excursions (MAGE) | 1 year
  MAGE is measured by applying continuous glucose monitoring system (CGMS) on subjects in each follow-up of this one-year study.

SECONDARY OUTCOMES:
Change in HbA1C | 1 year
Change in C-peptide | 1 year
Change in insulin dose | 1 year
  hyperglycemic and hypoglycemic events.
Hyperglycemic and hypoglycemic events | 1 year
  Blood sugar level higher than 11.1 mmol/l or lower than 3.9 mmol/l.
Life quality evaluation | 1 year
  Number of subjects with disturbance of emotion, sleep, resting or energy.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Rondas D, D'Hertog W, Overbergh L, Mathieu C. Glucagon-like peptide-1: modulator of beta-cell dysfunction and death. Diabetes Obes Metab. 2013 Sep;15 Suppl 3:185-92. doi: 10.1111/dom.12165. PMID 24003936
- [Background] Chang TJ, Tseng HC, Liu MW, Chang YC, Hsieh ML, Chuang LM. Glucagon-like peptide-1 prevents methylglyoxal-induced apoptosis of beta cells through improving mitochondrial function and suppressing prolonged AMPK activation. Sci Rep. 2016 Mar 21;6:23403. doi: 10.1038/srep23403. PMID 26997114
- [Background] Mathieu C, Gillard P. Arresting type 1 diabetes after diagnosis: GAD is not enough. Lancet. 2011 Jul 23;378(9788):291-2. doi: 10.1016/S0140-6736(11)60978-1. Epub 2011 Jun 27. No abstract available. PMID 21715000